CLINICAL TRIAL: NCT00656240
Title: A Randomized, Double-Masked, Parallel-Group Trial of DE-104 Ophthalmic Solution in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: To Investigate the Safety and Efficacy of DE-104 Ophthalmic Solution to Treat Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Other Study IDs: 01040703
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: DE-104 ophthalmic solution
- 2 (Experimental)
  Interventions: Drug: DE-104 vehicle

INTERVENTIONS:
Drug: DE-104 ophthalmic solution
  Arms: 1
Drug: DE-104 vehicle
  Arms: 2

SUMMARY:
To investigate the intraocular pressure (IOP)-lowering effect and safety of DE-104 ophthalmic solution in patients with Primary Open-Angle Glaucoma or Ocular Hypertension

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open-angle glaucoma or ocular hypertension.
* Provided signed, written informed consent.
* If a subject is a female of childbearing potential, she must utilize reliable contraceptive throughout the study, and must have a negative urine pregnancy test prior to enrollment into this study.

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy, or females of childbearing potential who are not using a reliable method of contraception.
* Presence of any abnormality or significant illness that could be expected to interfere with the study.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka, Japan, Osaka, Japan